CLINICAL TRIAL: NCT03065842
Title: A Pre and Post Test Intervention Program to Prevent Abortion and Contraceptive-use Stigma Among School Youths in Kenya: A Quasi-Experimental Design
Brief Title: A Pre and Post Test Intervention Design to Prevent Abortion and Contraceptive-use Stigma Among School Youths in Kenya
Acronym: SAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: University of Nairobi (Other); Moi University (Other)
Responsible Party: Principal Investigator, Marlene Makenzius, Principal Investigator, RNM, MPH, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4-3163/2015
Record Dates: First submitted 2017-02-17; First posted 2017-02-28 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Social Stigma; Pregnancy; Contraception
Keywords: Stigma; Pregnancy; Abortion; Contraception; Adolescence
MeSH Terms: conditions — Social Stigma | interventions — Abortion, Induced

STUDY DESIGN:
Intervention Model Description: A quasi-experimental design, which is the Comparison Group Pre-test/Post-test Design, as in the current design. This design is the same as the classic controlled experimental design except that the subjects cannot be randomly assigned to either the experimental or the control group. The design came out because of difficulty of applying the classical natural science method to the social or the researcher cannot control which group will get the treatment, for example interventions targeting school students.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abortion- and contraceptive-use stigma reduction program (Experimental): Four sessions (à 120 min), every week in 1 month.
  Interventions: Behavioral: Abortion- and contraceptive-use stigma reduction program
- Usual standards (Active Comparator): Usual standards
  Interventions: Behavioral: Usual Standards

INTERVENTIONS:
Behavioral: Abortion- and contraceptive-use stigma reduction program — An abortion- and contraceptive-use stigma reduction intervention (3-weeks), capturing i. Negative stereotypes associated with girls who have had an abortion. ii. Discrimination/exclusion of girls who have had an abortion. iii. Fear of coming in contact with a girls who have had an abortion. iv. Negative stereotypes about girls using a contraceptive method. v. Misconceptions about contraceptive use.
  The pedagogy will be based on that gender stereotypes, intent to control female sexuality, compulsory motherhood, are social constructs that can be deconstructed. Pedagogical methods will include role modelling, practice of desired behaviours, activities for building self-efficacy, and didactic instructions.
  Other Names: SAC - Stigma Abortion Contraception
  Arms: Abortion- and contraceptive-use stigma reduction program
Behavioral: Usual Standards — Usual standards according to the school curriculum in Kenya.
  Arms: Usual standards

SUMMARY:
In many low-income countries, unsafe abortion is recognized as a leading cause of maternal morbidity and mortality. Social stigma surrounding abortion and contraceptive use plays a critical role in the social, medical, and legal marginalization of abortion and contraceptive services. Though this stigma is pervasive and threatens women's health, it is not well understood how it can be reduced. The Stigmatizing Attitudes, Beliefs and Actions Scale (SABAS) was designed in 2013, to measure abortion stigma at individual and community level. Objective: I) to conceptualize abortion stigma among; health care providers, secondary school teachers and students, and II) to determine if a school based intervention targeting stigma specifically faced by girls when accessing abortion and contraceptive services, compared to usual standards, will decrease related stigma and increase contraceptive use among students, who are sexually active. Design, Setting, Participants: I) Focus group discussions (FGD) with service providers at YFC (n=12), secondary school teachers (n=16) and secondary school students (n=20), and II) a quasi-experimental pre- and post-intervention study, targeting 800 secondary school students (14-20 y), in Kisumu, Kenya. Two schools will be assigned; one interventions unit (n=400 students) and one control unit (n=400 students). The schools are similar according to the study site, size and academic standards. The region is chosen because of its low rate of contraceptive use, and high rate of teen pregnancy and of unsafe abortions. Standard deviation is the measure of dispersion or variability in the data. The sample size of 400 is based on a previous study and will give a power of 80% to detect differences (95% Cl) between the two groups. Intervention: An abortion- and contraceptive-use stigma reduction intervention (1-month program), capturing negative stereotypes about women that are associated with abortion and contraceptive use. Main Outcome: Abortion-stigma reduction. Secondary outcome: Contraceptive-use stigma reduction. Measured at baseline (pre-test), and post-test at 1- and 12-months, by using the validated SABA-scale. Analyses: Qualitative content analysis and repeated measures, ANOVA.

Funded by: The Swedish Research Council for Health, Working Life and Welfare 2015-01194, and The Swedish Research Council 2016-05670

DETAILED DESCRIPTION:
Today, abortion is one of the most common practices within gynaecological care. Despite its existence across time and its persistence across geographic location, the impact of abortion on women, families, communities and societies differs a lot across the world. Safe abortions - done by trained providers in hygienic settings and particularly early medical abortions carry fewer health risks. In countries like Sweden, Romania, Nepal and South Africa, liberalisation of abortion laws has had a direct and positive impact on maternal mortality. Yet, approximately half of the 42 million abortions that take place every year are unsafe. Nearly one in five maternal deaths can be attributed to unsafe abortion, and more than 500 women per 100,000 live births die from consequences of unsafe abortions. There is an inherent need to invest in intervention strategies to improve maternal health, especially amongst youth.

Until recently, abortion was only legally permissible in Kenya to save the life of a woman, but a new constitution adopted in 2010 makes abortion available to protect a woman's health. Article 43 in the constitution further widens access to reproductive health rights, as every person has the right to the highest attainable standard of health, which includes the right to health care services, including reproductive health care. However, contraceptive use remains low in Kenya. Consequently unwanted pregnancy and unsafe abortions are common, many of which require medical care for complications. A Kenyan woman has a one in 55 chance of dying from pregnancy related causes over her lifetime, and about 360 women per 100,000 live births die.

Sexuality education is part of general education. Its preventive nature not only contributes to the prevention of negative consequences linked to sexuality, but can also improve quality of life, health and well-being. In this way, sexuality education contributes to health promotion in general. In some countries SRE in school is compulsory, as for example in Sweden. In Kenya, SRE is not compulsory in the teacher education. Many teachers receive additional training, although this training has a focus on teaching about HIV/AIDS. Oginga (2014) recommend that SRE need to be incorporated and compulsory in the teacher-training curriculum in Kenya.

While extensive research has investigated the public health consequences of unwanted pregnancy and unsafe abortion from a human rights perspective, there is little research on stigma related to contraceptive use and abortion among youths. Causes of abortion stigma such as negative gender stereotypes, intent to control female sexuality, compulsory motherhood - are social constructs that can be deconstructed. Women's subordinate status in most societies has negative implications for women's sexual and reproductive health and rights (SRHR).

Although there is lack of research on stigma related to contraceptive use and abortion and how it can be reduced, the occurrence of such stigma are widely acknowledged in many countries. Few conceptual and methodological tools exist to measure its effects. For many years now, the International Planned Parenthood Federation (IPPF), together with partner organizations, has implemented programmes to specifically address and combatting HIV stigma. In the past five years there has been increased global attention on abortion stigma. IPPF has thus expanded its work to address the impact that negative beliefs and attitudes about abortion has on access to, and scale-up of, safe abortion services. Abortion stigma manifests at many levels, from individuals and service providers to communities, institutions, laws and policies, and wider public discourse including the media.

In 2013, Ipas developed a scale to measure abortion stigma at the individual and community levels, the Stigmatizing Attitudes, Beliefs and Actions Scale (SABAS), to inform the development of interventions to mitigate stigma.

PROJECT DESCRIPTION Purpose and Aims

This project has mixed-methods approach, a qualitative and quantitative quasi-experimental pre- and post-intervention design. The purpose is to empirically determine what role stigma related to abortion and contraceptive use plays, how it is expressed, and how it can be countered most effectively.

Firstly, the aim is to conceptualize abortion stigma, among health care providers in YFC, and among teachers and students in secondary schools. Secondly, to determine if a school based intervention, compared to usual standards, will decrease abortion- and contraceptive-use stigma and increase contraceptive use among sexually active secondary school students.

METHODOLOGY The social and political sensitivity surrounding induced abortion makes it very difficult to conduct high-quality research to measure its incidence and related stigma, which automatically introduces bias into the result. Surveys of providers are also problematic for a number of reasons, as for example in countries where safe abortion is illegal for obvious reasons (fear of prosecution). Therefore the investigators have chosen to use qualitative- and quantitative approaches (data triangulation) to conceptualize abortion and contraceptive use stigma, and to estimate and validate the incidence.

Design: I) a qualitative approach with Focus Group Discussions (FGDs), and II) a quantitative quasi-experimental pre- and post-intervention study design, comparing student attitudes in intervention schools and matched control schools will be used. Tool: SABA-scale will be used to assess attitudes and behaviour at baseline (pre-test) and post-test at 1 and 12 month. Primary out outcome: Abortion-stigma. Secondary outcome: Contraceptive-use stigma.

Settings: Potential schools in semi-urban settlements in the county of Kisumu, will be identified according to the study site, size and academic standards (public schools). The schools will be ordered alphabetically by name and imported into a statistical computer software by an IT-assistant at Kisumu Medical and Educational Trust (KMET), Kisumu. The software will randomly generate the allocation schedule for assignment of the stigma reduction intervention to one school, and one to be operated as a control school. This area has a dominance of Christian religions, Luo, Luhya and Kisii ethnic groups, and low socio-economic status (SES) reflect the regional profile.

Participants: I) Service providers (n=12) in YFC, secondary school teachers (n=16) and will participate in gender mixed FGDs, and students (females, n=10; males, n=10), and II) secondary school students between 14 and 20 years (n=200 male students; 200 female students), will be included in the intervention unit, and the about the same number in the control unit.

Measurements: The Stigmatizing Attitudes, Beliefs and Actions Scale (SABAS) is a tool designed to measure abortion stigma at the individual and community level. A 57-item instrument was created in 2013, pre-tested, and administered to 531 individuals (n=250 in Ghana and n=281 in Zambia). All analyses were completed using Stata IC/11.2. SABAS captures three important dimensions of abortion stigma: negative stereotypes (8 items), discrimination and exclusion (7 items), and potential contagion (3 items) (1). IPPF adapted the Stigmatising Attitude, Beliefs and Actions Scale (SABAS) developed by Ipas to measure abortion stigma amongst community members in the project areas in Benin, Burkina Faso, India and Pakistan at the outset and end of the Packard Foundation abortion stigma project 2014-2016. The response categories in SABAS have a Likert format from "strongly disagree" to "strongly agree" with each response being assigned a value ranging from 1-5. The tool can be used in several ways: for example as baseline and/or endline data collection in stigma-reduction interventions or as a "pre and post-test" to measure short-term change at the individual and/or community level. The SABA tool will be further modified to adapt the tool to the context of this setting. In addition new questions will be drafted targeting gender stereotypes related to girls and contraceptive-use and misconceptions (including condom use) at last sexual intercourse (yes/no). These questions will be drafted in collaboration with providers, teachers and students, study I (FGD). This adapted tool will be used at baseline (pre-test) and post-test at 1 and 12 months, to measure short- and long-term change at both group- and individual level.

Analysis and sample size calculation: Study I) data will be qualitatively analysed according to guide for exploring contraceptive- and abortion-related stigma. Study II). The sample size will take into account to identify a 25% stigma reduction (one-sided t-test), using a 95% CI (α=0.05). The sample size was preliminary calculated to be about 1,200 and arbitrarily derived since the 2 schools were drawn from a regional sample frame of four gender-mixed christian schools with a minimum of 400 students (similar schools according to study site, SES, and academic standards). However, for the initial validation of the scales the sample size (n = 300/school) was based on the principle of a minimum of ten respondents (5/gender) per scale item, and with a drop-out rate of 20%, and a further loss to follow-up of the final-year students who participated in the intervention but were not planned to be followed up at one-year, as they will have left the school (~30%).

The outcome of the intervention will be analysed quantitatively according to Shellenberg et al (2013). A higher score on the SABAS represents more stigmatizing attitudes and beliefs. There is no predetermined cut-off or threshold for what represents stigma. The results will guide us if to use the scores as continuous variables or to create cut-offs that are appropriate to the context/setting. For continuous variables, the intervention effect are to be analyzed using repeated measures ANOVA (PASW 20.0), significant p-value >0.05. Within-subjects factor: time. Between-subjects factor: intervention vs. control. Dependent variable: SABAS attitudes, beliefs and actions items.

ETHICAL CONSIDERATIONS Ethical clearance is recieved from JOOTRH/CDC in Kisumu, research and ethics authority who will review the proposal for approval before the project starts. All participants will be asked to give a written consent. For participants who are below 18 years, we will obtain parental consent as well as approval from the Ministry of education. Consent forms will be translated into Kiswahili language and back translated into English to ensure accurate translation. The participants will be informed that they can withdraw from participation at any time without any consequences. The research team will ensure that all research data, regardless of format, is stored securely and backed up or copied regularly. All data will be handled according to national laws and guidelines. Prof Edwin Were, a research team member is also a member in a regional ethical committee, and he will overview the ethical aspects in this study, in accordance to national laws and guidelines.

PROJECT TEAM AND COLLABORATORS Professor Kristina Gemzell-Danielsson, Karolinska University Hospital, head of the research group at the WHO-collaborating centre at the department of Obstetrics and Gynaecology, Karolinska Institutet has extensive experiences from conducting international randomised control trials within Human Reproduction. Professor Elisabeth Faxelid, Karolinska Institutet and Associated professor Marie Klingberg-Allvin, Högskolan Dalarna has long experiences of international intervention- and facility-based research. The applicant, Marlene Makenzius, has previous experiences from research related to induced abortion among Swedish women and men (Uppsala University), Public Health Policy analyses at a national level (The National Agency of Public Health, Sweden), practical work as midwife at YFC and have currently monitored a post-abortion care project in Kisumu (RCT-study).

The following Kenyan researchers will be involved in the project: Monica Oguttu, PhD RNM, Head of KMET, Sam Owoko, Program manager at KMET, currently involved in a male-involvement project and a STI/HIV-intervention in primary schools, Dr. Paul Mitei Obs/Gyn practitioner and traiinig expert with vast experience and also involved in PAC study, currently KCH Obs/Gyn. Caroline Nyandat, Midwife/nurse, Coordinator at KMET, currently involved quality development in a YFC, Edwin Were, is professor of Reproductive Health at Moi University in Eldoret, with long experience in clinical service provision and managing clinical trials and also serves in a local ethics committee. Theresa Mary Awuor, nurse midwife, BscN, a PhD student, experience in leadership currently a member of the Technical working Group-Global Health Leadership with a consortium of universities in the United States of America and African Universities called Afya Bora, and Beatrice Otieno, data clerk at KMET.

PRINCIPLE INVESTIGATORS Marlene Makenzius from Sweden and Monica Oguttu from Kenya.

SIGNIFICANCE IN KENYA The complications from unsafe abortion continue to pose a serious threat to Kenyan women's health. Nearly 120,000 women received care in health facilities for complications resulting from unsafe abortions in 2012, corresponding to an induced abortion ratio of 30 abortions per 100 births in 2012. Severe complications of unsafe abortions were most common among women aged 10-19. More than 70% of women seeking post-abortion care were not using a method of contraception prior to becoming pregnant. The investigators believe that the potential benefit of this study is high on a community level as well as the individual level. The participants may also benefit as the intervention targets contraceptive use and may thus reduce unwanted pregnancy. Unwanted pregnancy undermines young peoples' (especially women's) schooling, health, social status and future opportunities for work. Young people will therefore benefit from reduced abortion-stigma and increased contraceptive use. In addition, in Kisumu this study will

* Encourage SRH as part of the regular curriculum in secondary schools.
* Encourage male involvement in health-seeking practices and women's reproductive health.
* Increase access to contraceptive-use among students .
* Identify and empower representatives from the communities; school- and church leaders, and open meetings for publics (Baraza), to sensitize and influence communities on problems of unsafe abortion and low contraceptive use.
* Establishment of environments and capacity among international, national and regional research actors and leading NGO's to mitigate the gap between knowledge and practice in the prevention of unsafe abortions.
* Enable women within the project to undergo research training that will facilitate development of local and regional academic competence.
* Create awareness of gender equality perspective in research.

ELIGIBILITY:
Inclusion Criteria:

* Secondary school students between 14 and 20 years

Exclusion Criteria:

* Age below 14 years

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1207 (Actual)
Dates: Start 2017-02-05 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
Stigmatizing attitudes associated with girls who have had an abortion: To assess a reduction from baseline attitudes at 12 months | Baseline, and post-test at 12 months
  Measured with the SABA-scale

SECONDARY OUTCOMES:
Stigmatizing attitudes associated with girls using a contraceptive method: To assess a reduction from baseline attitudes at 12 months | baseline, and post-test at 12 month
  Measured with a questionnaire (likert scale)
Stigmatizing attitudes associated with girls who have had an abortion: To assess a reduction from baseline attitudes at 1 month | baseline, and post-test at 1 month
  Measured with the SABA-scale
Stigmatizing attitudes associated with girls using a contraceptive method: To assess a reduction from baseline attitudes at 1 month | baseline, and post-test at 1 month
  Measured with a questionnaire (likert scale)

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Makenzius, PhD, Principal Investigator — Karolinska Institutet; Monica Oguttu, PhD, Principal Investigator — Kisumu Medical Education Trust, Kenya
Locations (1):
- Secondary schools in Kisumu, Kisumu, Kisumu County, Kenya

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shellenberg KM, Hessini L, Levandowski BA. Developing a scale to measure stigmatizing attitudes and beliefs about women who have abortions: results from Ghana and Zambia. Women Health. 2014;54(7):599-616. doi: 10.1080/03630242.2014.919982. PMID 25074064
- [Background] Makenzius M, Tyden T, Darj E, Larsson M. Repeat induced abortion - a matter of individual behaviour or societal factors? A cross-sectional study among Swedish women. Eur J Contracept Reprod Health Care. 2011 Oct;16(5):369-77. doi: 10.3109/13625187.2011.595520. Epub 2011 Jul 21. PMID 21777046
- [Background] Makenzius M, Tyden T, Darj E, Larsson M. Women and men's satisfaction with care related to induced abortion. Eur J Contracept Reprod Health Care. 2012 Aug;17(4):260-9. doi: 10.3109/13625187.2012.688149. Epub 2012 Jul 3. PMID 22758772
- [Background] Makenzius M, Tyden T, Darj E, Larsson M. [Sweden has the highest abortion rate among the Nordic countries. Unwanted pregnancies should be seen in a holistic perspective--individuals, health care, community]. Lakartidningen. 2013 Sep 18-24;110(38):1658-61. No abstract available. Swedish. PMID 24199440
- [Background] Sedgh G, Singh S, Shah IH, Ahman E, Henshaw SK, Bankole A. Induced abortion: incidence and trends worldwide from 1995 to 2008. Lancet. 2012 Feb 18;379(9816):625-32. doi: 10.1016/S0140-6736(11)61786-8. Epub 2012 Jan 19. PMID 22264435
- [Background] Grimes DA, Benson J, Singh S, Romero M, Ganatra B, Okonofua FE, Shah IH. Unsafe abortion: the preventable pandemic. Lancet. 2006 Nov 25;368(9550):1908-19. doi: 10.1016/S0140-6736(06)69481-6. PMID 17126724
- [Background] Hord C, David HP, Donnay F, Wolf M. Reproductive health in Romania: reversing the Ceausescu legacy. Stud Fam Plann. 1991 Jul-Aug;22(4):231-40. PMID 1949105
- [Background] Jewkes R, Rees H. Dramatic decline in abortion mortality due to the Choice on Termination of Pregnancy Act. S Afr Med J. 2005 Apr;95(4):250. No abstract available. PMID 15889846
- [Background] Swedish National Institute of Public Health [SNIPH]. Sexualitet och reproduktiv hälsa. Kunskapsunderlag för Folkhälsopolitisk rapport 2010 [Sexuality and reproductive health. Public health report 2010] Östersund2011 [cited 2016 12 Februari]. Available from: https://www.folkhalsomyndigheten.se/pagefiles/12538/R2011-02-Sexualitet-och-reproduktiv-halsa.pdf
- [Background] Henderson JT, Puri M, Blum M, Harper CC, Rana A, Gurung G, Pradhan N, Regmi K, Malla K, Sharma S, Grossman D, Bajracharya L, Satyal I, Acharya S, Lamichhane P, Darney PD. Effects of abortion legalization in Nepal, 2001-2010. PLoS One. 2013 May 31;8(5):e64775. doi: 10.1371/journal.pone.0064775. Print 2013. PMID 23741391
- [Background] National Council for Law Reporting. Constitution of Kenya 2010. National Council for Law Reporting with the Authority of the Attorney-General.
- [Background] Makenzius M, Larsson M. Early onset of sexual intercourse is an indicator for hazardous lifestyle and problematic life situation. Scand J Caring Sci. 2013 Mar;27(1):20-6. doi: 10.1111/j.1471-6712.2012.00989.x. Epub 2012 Mar 28. PMID 22462801
- [Background] Makenzius M, Gadin KG, Tyden T, Romild U, Larsson M. Male students' behaviour, knowledge, attitudes, and needs in sexual and reproductive health matters. Eur J Contracept Reprod Health Care. 2009 Aug;14(4):268-76. doi: 10.1080/13625180903015871. PMID 19526422
- [Background] World Health Organization W. Europe and BZgA Standards for Sexuality Education in Europe. A framework for policy makers, educational and health authorities and specialists. Cologne: Federal Centre for Health Education, BZgA 2010.
- [Background] Oginga EA. The Factors Influencing The Teaching Of HIV/AIDS Education In Public Primary Schools In Kisumu East. Int J of Education and Research. 2014;2(1).
- [Background] Makenzius M, Tyden T, Darj E, Larsson M. Risk factors among men who have repeated experience of being the partner of a woman who requests an induced abortion. Scand J Public Health. 2012 Mar;40(2):211-6. doi: 10.1177/1403494811435496. Epub 2012 Feb 3. PMID 22307996
- [Background] Shellenberg KM, Moore AM, Bankole A, Juarez F, Omideyi AK, Palomino N, Sathar Z, Singh S, Tsui AO. Social stigma and disclosure about induced abortion: results from an exploratory study. Glob Public Health. 2011;6 Suppl 1:S111-25. doi: 10.1080/17441692.2011.594072. Epub 2011 Jul 11. PMID 21745033
- [Background] Wellings K, Jones KG, Mercer CH, Tanton C, Clifton S, Datta J, Copas AJ, Erens B, Gibson LJ, Macdowall W, Sonnenberg P, Phelps A, Johnson AM. The prevalence of unplanned pregnancy and associated factors in Britain: findings from the third National Survey of Sexual Attitudes and Lifestyles (Natsal-3). Lancet. 2013 Nov 30;382(9907):1807-16. doi: 10.1016/S0140-6736(13)62071-1. Epub 2013 Nov 26. PMID 24286786
- [Background] Makenzius M, Tyden T, Darj E, Larsson M. Autonomy and dependence--experiences of home abortion, contraception and prevention. Scand J Caring Sci. 2013 Sep;27(3):569-79. doi: 10.1111/j.1471-6712.2012.01068.x. Epub 2012 Aug 22. PMID 22913927
- [Background] Kumar A, Hessini L, Mitchell EM. Conceptualising abortion stigma. Cult Health Sex. 2009 Aug;11(6):625-39. doi: 10.1080/13691050902842741. PMID 19437175
- [Background] Shellenberg KM, Tsui AO. Correlates of perceived and internalized stigma among abortion patients in the USA: an exploration by race and Hispanic ethnicity. Int J Gynaecol Obstet. 2012 Sep;118 Suppl 2:S152-9. doi: 10.1016/S0020-7292(12)60015-0. PMID 22920620
- [Background] Onyango MA, Owoko S, Oguttu M. Factors that influence male involvement in sexual and reproductive health in western Kenya: a qualitative study. Afr J Reprod Health. 2010 Dec;14(4 Spec no.):32-42. PMID 21812196
- [Background] Greene M, Mehta M, Pulerwitz J, Wulf D, Bankole A, Singh S. (2010),.Involving Men in Reproductive Health: Contributions to Development. MillenniumProject. UN. 2010.
- [Background] Billings D, Hessini L, Andersen K. (2016) Focus group guide for exploring abortion-related stigma. Chapel Hill, NC: Ipas: 2009. International Parenthood Federation. Addressing abortion stigma. IPPF, UK,. [cited 2016 25 May]. Available from: http://www.ippf.org/resource/Addressing-abortion-stigma
- [Background] Bandura A. Ontological and epistemological terrains revisited. J Behav Ther Exp Psychiatry. 1996 Dec;27(4):323-45. doi: 10.1016/s0005-7916(96)00049-3. PMID 9120037
- [Background] Singh S, Remez L, Tartaglione A, eds (2004). Methodologies for Estimating Abortion Incidence and Abortion-Related Morbidity: A Review. New York: Guttmacher Institute and Paris International Union for the Scientific Study of Population, 2010. Research Methods, Instruments, & Computers; 32(2): 347-356.
- [Background] Graneheim UH, Lundman B. Qualitative content analysis in nursing research: concepts, procedures and measures to achieve trustworthiness. Nurse Educ Today. 2004 Feb;24(2):105-12. doi: 10.1016/j.nedt.2003.10.001. PMID 14769454
- [Background] Potvin PJ, Schutz RW. Statistical power for the two-factor repeated measures ANOVA. Behav Res Methods Instrum Comput. 2000 May;32(2):347-56. doi: 10.3758/bf03207805. PMID 10875184
- [Result] Ministry of Health. Incidence and Complications of Unsafe Abortion in Kenya - Key Findings of a National Study. The Republic of Kenya: Ministry of Health, 2013.
- [Derived] Hakansson M, Super S, Oguttu M, Makenzius M. Social judgments on abortion and contraceptive use: a mixed methods study among secondary school teachers and student peer-counsellors in western Kenya. BMC Public Health. 2020 Apr 15;20(1):493. doi: 10.1186/s12889-020-08578-9. PMID 32295574